CLINICAL TRIAL: NCT06627790
Title: Comparative Evaluation of Efficacy of a Potassium Nitrate Containing Herbal Mouthwash to a Potassium Oxalate Mouthwash in Dentinal Hypersensitivity - a Randomised Clinical Trial
Brief Title: Efficacy of a Potassium Nitrate Containing Herbal Mouthwash to a Potassium Oxalate Mouthwash in Dentinal Hypersensitivity
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. D. Y. Patil Dental College & Hospital (Other)
Collaborators: Jasberry Healthcare Pvt. Ltd (Unknown)
Responsible Party: Principal Investigator, D. Gopalakrishnan, DEAN PROFESSOR AND HOD, Dr. D. Y. Patil Dental College & Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DYPDCH/DPU/EC/582/130/2023
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Dentin Hypersensitivity
Keywords: dentinal hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Potassium nitrate containing herbal mouthwash (Experimental): Group A: Participants will be adviced to use mouthwash twice daily in 10ml volume for 60 seconds, 30 minutes after brushing and not to eat anything for 45 minutes
  Interventions: Drug: Mouthwash preparation
- Potassium oxalate mouthwash (Active Comparator): Group B: Participants will be adviced to use mouthwash twice daily in 10ml volume for 60 seconds, 30 minutes after brushing and not to eat anything for 45 minutes.
  Interventions: Drug: Mouthwash preparation

INTERVENTIONS:
Drug: Mouthwash preparation — Participants will be divided into two groups Group A and Group B Both the groups will receive thorough scaling and root planing at required sites. Use of mouthwash preparation is adviced for 8 weeks and discontinue after for 4 weeks. The Visual analogue scale Hypersensitivity will be assessed via Visual Analogue Scale at 4, 8 and 12 week interval

SUMMARY:
The goal of this clinical trial is to compare the efficacy of potassium nitrate containing herbal mouthwash to potassium oxalate mouthwash in management of dentinal hypersensitivity.

* Participants will be divided into two groups by computer generated randomization. The participants will be divided into two groups, Group 'A' and Group 'B' by Simple Random Allocation as both groups, each group will involve 20 participants with at least two sites showing dentinal hypersensitivity
* The assessment of Dentinal Hypersensitivity will be done after scaling and/or root planing (if required) by subjecting affected sites with Air Blast Test (ABT), Cold Water Test (CWT) and Tactile Response assessment will be recorded using Visual Analogue Scale (VAS). All sensitivity tests will be executed by a single examiner who will be blinded to the randomization and will record DH at baseline and at 4, 8 and 12 weeks

DETAILED DESCRIPTION:
Mouthwash has become accepted as a preferable delivery vehicle compared to pastes and gels due to ease of their use and access to all the areas of the mouth and ability to circumvent the discomfort that could occur when brushing the sensitive dentin surface because the osmolarity of toothpaste may increase pain sensations.

This clinical trial is designed to assess the clinical efficacy of a Potassium nitrate containing Herbal mouthwash (Jasmate Klinika Mouthwash) compared with Potassium oxalate containing mouthwash (Listerine Advance Defense Sensitive Mouthwash). The Jasmate Klinika Mouthwash contains Curcumin and Potassium Nitrate as active ingredients. The concentration of Potassium Nitrate (KN) is 5% and Curcumin is 2%. The Listerine Advance Defense Sensitive Mouthwash contains Potassium Oxalate (KO) in 1.4% concentration.

* The participants will be divided into two groups, Group 'A' and Group 'B' by Simple Random Allocation as both groups, each group will involve 20 participants with at least two sites showing dentinal hypersensitivity
* The assessment of Dentinal Hypersensitivity will be done after scaling and/or root planing (if required) by subjecting affected sites with Air Blast Test (ABT), Cold Water Test (CWT) and Tactile Response assessment will be recorded using Visual Analogue Scale (VAS). All sensitivity tests will be executed by a single examiner who will be blinded to the randomization and will record DH at baseline and at 4, 8 and 12 weeks
* After the baseline assessment participants will be instructed for oral hygiene maintenance and the use of 10ml of mouthwash for rinsing twice daily for 60 seconds, 30 minutes after brushing the teeth with standard toothpaste and soft bristled toothbrush
* Participants will be asked to discontinue the use of mouthwash after 8 weeks and will be assessed at 12 weeks with Air Blast Test(ABT), Cold Water Test(CWT) and Tactile Response assessment will be done using Visual Analogue Scale(VAS)

ELIGIBILITY:
Inclusion Criteria:

* Participants with at least two DH sites with VAS score ≥4
* Participants with teeth showing cervical abrasion, erosion, gingival recession
* Participants >18 years in general good health
* Participants self-reporting with history of dentinal hypersensitivity to various stimuli.
* Participants with minimum 20 natural teeth

Exclusion Criteria:

* Teeth with severe caries, faulty restoration, prosthetic crown, chipping, fracture, symptoms of pulpal damage
* Participants who has taken long term analgesic therapy within 30 days before the start of the study
* Participants who have undergone any treatment for dentinal hypersensitivity in past 3 months
* Participants with ongoing orthodontic therapy
* Participants with history or presence kidney disorder, kidney stones, eating disorders, uncontrolled gastro-oesophageal reflux disease, excessive exposure to acids or any other systemic condition that predisposes to dentinal hypersensitivity
* Severe Periodontal disease characterized by extensive tooth mobility and or extensive alveolar bone loss involving 10 or more teeth
* Women who are pregnant or lactating

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Dentinal Hypersensitivity | at 4, 8 and 12 week interval
  The dentinal hypersensitivity will be assessed using Visual Analogue Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. D Y Patil dental College and Hospital, Pimpri, Pune, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No